CLINICAL TRIAL: NCT02758938
Title: End User Assessment of Urological Biofeedback Game Software
Brief Title: Urological Biofeedback Game Software
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2015-0235
Record Dates: First submitted 2015-12-29; First posted 2016-05-03 (Estimated); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Lower Urinary Tract Symptoms
MeSH Terms: conditions — Lower Urinary Tract Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Patient Subjects (Experimental): Patients that are part of the UW LUTD Program (n=30) will undergo 3 weekly biofeedback sessions each lasting 1 hour. All interactive biofeedback sessions will be conducted by American Family Children's Hospital nurses that are experienced in standard biofeedback techniques. After the patient has completed all of the biofeedback sessions, he/she will complete a feedback form about their satisfaction with the device.
  Interventions: Other: Urologic biofeedback software
- Biofeedback Nurse Subjects (Experimental): The nurses (n=3) involved in the biofeedback portion of the UW LUTD Program will undergo a Nurse Training Session where they will be asked to "think aloud" while completing an outlined scenario. Their feedback will be used to update the software to make it more user friendly. After the session, they will be asked to complete the System Usability Scale (SUS). Additionally, after guiding patients through biofeedback sessions using the new software, they will be asked to complete the Nurse Feedback Form.
  Interventions: Other: Urologic biofeedback software
- Biofeedback Physician Subject (Experimental): The physician (n=1) that oversees the UW LUTD Program will assess data from each patients session. Based on the information he gathers from the session, he will complete a feedback form. Each patient's EMG activity will be stored by the video game which will allow the physician to review the patient's performance. Specifically, the physician will look for the minimum relaxation and the maximum contraction levels of the patient throughout play as well as muscular isolation.
  Interventions: Other: Urologic biofeedback software
- Focus Group Subjects (Experimental): A Focus Group session will involve the physician involved in this study, an advisor on the project and staff involved in the project as well as three random individuals outside of the project (n=7). These individuals will provide feedback on the software that will be used to improve the software.
  Interventions: Other: Urologic biofeedback software

INTERVENTIONS:
Other: Urologic biofeedback software — All subjects (end users) will be walked through the urologic biofeedback software training suite. Each end user will follow a protocol that is specific to their role. Upon completing their session(s) with the software, each end user will provide appropriate feedback.

SUMMARY:
The goal of this study is to test the usability of updated biofeedback game software developed to help train the muscles involved in lower urinary tract dysfunction (LUTD) through electromyography (EMG) controlled video games.

A Windows-DOS based biofeedback game system is currently used at the investigator's institution to help treat LUTD in pediatric patients. This system, however, is outdated and needs to be replaced with updated hardware and software. A new updated system was recently created by University of Wisconsin-Madison (UW) Biomedical Engineering students. This system utilizes a FDA approved EMG device (SRS Medical Aware™ EMG Dual Muscle Monitor) paired with biofeedback game software that was developed by the students. The investigators wish to test the usability of the new software to identify areas that need improvement to make the software more user-friendly.

This study will evaluate the end users' (i.e., physician, biofeedback nurses, patients) perception of the updated software. In determining usability, we hope to 1) decrease risk of end user error; 2) make the software intuitive (easier to use); 3) decrease reliance on the user manual; 4) decrease need for training; and 5) increase understanding of software operation. This will be an ongoing study in which we continuously monitor the usability of the software as it is updated based on end-user feedback. The investigators plan to do all usability testing under the same IRB protocol. If further testing involves items not discussed here, a "new change" will be made to the IRB application.

DETAILED DESCRIPTION:
BACKGROUND AND SIGNIFICANCE

Medical and Biological:

LUTD is a common problem in children that can result in wetting during the day and night, frequent and urgent urination and urinary tract infections. In a subset of children, LUTD is the result of dis-coordination between pelvic floor and abdominal muscles. These children tend to contract their pelvic muscles rather than relax them during voiding. This abnormal contraction results in bladder changes that can result in incontinence. In most cases, understanding how to contract and relax the pelvic floor and abdominal muscles can help reduce LUTD symptoms. Identifying and learning how to utilize the pelvic floor without abdominal muscle activation is one of the most powerful effectors of bladder function.

The current LUTD Program at the investigator's institution includes a full history and physical exam followed by extensive education. If the patients do not improve they undergo additional evaluation with a renal pelvic ultrasound and simultaneous uroflowmetry and electromyography (EMG) study. Based on that evaluation a percentage of patients go on to receive biofeedback treatment. Biofeedback is typically recommended to patients who do not use the pelvic floor and abdominal muscles appropriately while voiding. The biofeedback treatment involves further education, standard biofeedback, and biofeedback computer games. In standard biofeedback, patients are made aware of their abdominal and pelvic floor muscle activity by a display that shows the abdominal and pelvic floor muscles' EMG activity. In the biofeedback computer games, patients control a variety of games with their pelvic floor and abdominal muscles. Both methods teach the patient how to locate the pelvic floor muscles and to isolate them while voiding. Biofeedback represents only one possible treatment plan for children with LUTD. Patients are analyzed prior to entering the biofeedback portion of the LUTD Program for compatibility with this treatment.

Several studies were conducted by McKenna and colleagues to assess the effectiveness of the biofeedback games on treating LUTD symptoms.The trials involved 41 and 160 children of varying ages that averaged out to be 7.2 and 8.5 years respectively. The games worked by acquiring feedback that represented a flexion of the pelvic floor and relaxation of the abdominal muscle. All of the children in the trials participated in approximately an hour of treatment per session that involved around 20 minutes of supervised gaming time. The 84% and 87% success rate in each trial showed that the method of using biofeedback paired with the video games is a viable option for the treatment of LUTD in children.

Motivation:

The investigator's institution has found success with using biofeedback games to train patients how to properly use their pelvic floor and abdominal muscles. Biofeedback is less invasive than traditional treatment methods and creates no potential harm to the patients. The DOS based biofeedback game system currently utilized at our institution is unique in that it involves the interaction of pelvic floor AND abdominal muscle to control video games through EMG signals. The system was created specifically for our LUTD Program and is not available on the market. The current biofeedback game system, however, has not been updated for almost 20 years and has become outdated. It requires a controller that is no longer available on the market, does not start reliably and overheats easily. Updated software and hardware are essential in order to keep this method of treatment available to the children at our institution.

Students from the UW Biomedical Engineering program created an updated biofeedback system to replace the current system. The system utilizes EMG hardware that has already been FDA approved paired with updated software created by the students. The device is still in the testing phase, but early consultation with the user population is necessary for assessing needs and developing requirements. Users also are critical for analytical work and testing throughout product development. The investigators plan to eventually market the software and field testing and feedback to manufacturers are highly desirable.

SPECIFIC AIMS/STUDY OBJECTIVES

Aims:

1. Evaluate physician's ability to read EMG values recorded throughout patient interaction with the software.
2. Evaluate the nurse reception of the new software, including usability of operation and setup.
3. Evaluate the patient's reception/satisfaction of the new video games that are part of the software package.

Outcomes:

Three metrics will be used to determine the usability of the video game software: 1) medical value to physician, 2) nurse ease of use, and 3) patient reception/satisfaction. Each of these metrics will be measured using evaluation forms specific to the role.

The goal is for the physicians and patients to rate usability at 50% or higher and for nurses to rate usability at 85 or higher (System Usability Score).

Because biofeedback uses well understood EMG technology, much of the system's success is related to patient satisfaction. Therefore, the first two aims seek to show usability in system setup and data presentation and our final aim will show usability according to patient engagement.

RESEARCH DESIGN AND METHODS

Study Population: A Focus Group session will involve the physician involved in this study, an advisor on the project and staff involved in the project as well as three random individuals outside of the project (7 total). These individuals will provide feedback on the software that will be used to improve the software. This study will also involve patients who are currently being treated in the UW LUTD Program under the supervision of Dr. Patrick McKenna. The investigators aim to recruit 30 of these patients who will complete the Patient Feedback Form. Additionally, the nurses (3 total) involved with biofeedback will provide qualitative and quantitative data in addition to completing the Nurse Feedback Form and the physician (1 total) involved with biofeedback will fill out the Physician Feedback Form.

Focus Group (Cognitive-Walk Through): To aid in the development of the final software to be used in the formal training below a set of informal peer focus group sessions will be held. These sessions will consist of Dr. Patrick McKenna, Christian Sauder, Joyce Jackson, Amit J. Nimunkar and three random individuals exterior to the project. During the session each participant will be asked to freely navigate through the training suite and game environment. During this activity they will be allowed to comment on the software and respond to follow up questions by the investigator. These questions and/or comments will be recorded by one of the investigators and used to guide the development process.

Nurse Training Session: After the Focus Group session, nurses will undergo a training session where qualitative and quantitative data on the software will be collected. The nurse will be asked to "think aloud" while completing an outlined scenario. Evaluators will be encouraged to vocalize their difficulties with the system and recommend changes to the interface design and functionalities. At the end of the think aloud session, an unstructured interview will be conducted during which user will be asked about their overall impression of the software and their suggestions for improving it. The think aloud session and unstructured interview will be recorded and transcribed by members of the study team. Each nurse will also be asked to complete the System Usability Scale (SUS).

Biofeedback: Upon delivering appropriate consent/assent forms, patients may begin biofeedback sessions with the new system. The patients will undergo 3 weekly sessions each lasting 1 hour. At each session, patients will have EMG-surface electrode patches (Kendall, 1050NPSM Neonatal Electrodes-Prewired, Small Cloth) placed at the 3 and 9 o'clock positions on the perineum to measure electrical activity of the pelvic floor muscle group. An additional surface electrode patch will be placed on the rectus abdominus to measure abdominal muscle activity. All interactive biofeedback testing will be conducted by American Family Children's Hospital nurses that are experienced in standard biofeedback techniques.

End User Assessment Forms: After the patient has completed all of the biofeedback sessions, he/she will complete a feedback form about their satisfaction with the games. The physician will complete a feedback form that assesses the medical value of the device and the nurses will complete a feedback form that assesses the ease of use of the device.

ELIGIBILITY:
Inclusion Criteria for Peer Focus Group:

• >18 years old

Inclusion Criteria for Patients:

* 6-18 years of age
* Diagnosed with LUTD
* Currently undergoing biofeedback in the UW LUTD Program

Exclusion Criteria for Patients:

* Patients who cannot complete the 6-week training program
* Patients receiving other treatment methods for LUTD throughout the program

Inclusion Criteria for Nurses (no exclusion criteria):

• Currently conducting biofeedback treatment in the UW LUTD Program

Inclusion Criteria for Physician (no exclusion criteria):

• Oversees biofeedback treatment and the UW LUTD Program

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-06; Primary Completion 2018-01 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Physician Feedback Form | 15 minutes
  This survey will measure the medical value that the software provides to the physician. The physician will be asked to rate certain items on a scale of 1 to 5 - 1 indicating "strongly agree" and 5 indicating "strongly disagree". Each item must score a 4 or 5 for the software to be considered "usable".
Nurse Feedback Form | 15 minutes
  This survey will identify the software's "ease of use" for the nurse. The nurses will be asked to rate certain items on a scale of 1 to 5 - 1 indicating "strongly agree" and 5 indicating "strongly disagree". Each item must score a 4 or 5 for the software to be considered "usable".
Patient Feedback Form | 15 minutes
  This survey will identify the patient's satisfaction with the software. The patients will be asked to rate certain items on a scale of 1 to 5 - 1 indicating "strongly agree" and 5 indicating "strongly disagree". Each item must score a 4 or 5 for the software to be considered "usable".
System Usability Scale (SUS) | 15 minutes
  This is a validated survey that measures that software's usability. Usability will be defined as a SUS score greater than or equal to 85 (Orfanou et al. 2015).

CONTACTS AND LOCATIONS:
Locations (1):
- American Family Children's Hospital, Madison, Wisconsin, United States

REFERENCES:
- [Background] McKenna PH, Herndon CD, Connery S, Ferrer FA. Pelvic floor muscle retraining for pediatric voiding dysfunction using interactive computer games. J Urol. 1999 Sep;162(3 Pt 2):1056-62; discussion 1062-3. doi: 10.1016/S0022-5347(01)68065-0. PMID 10458431
- [Background] Herndon CD, Decambre M, McKenna PH. Interactive computer games for treatment of pelvic floor dysfunction. J Urol. 2001 Nov;166(5):1893-8. PMID 11586256
- See also: Sawyer D. Do It By Design: An Introduction to Human Factors in Medical Devices 1996 — https://elsmar.com/pdf_files/FDA_files/DOITPDF.PDF
- See also: Orfanou et al. Perceived Usability Evaluation of Learning Management Systems: Empirical Evaluation of the System Usability Scale 2015 — http://www.irrodl.org/index.php/irrodl/article/view/1955/3262